CLINICAL TRIAL: NCT02887040
Title: A Randomized Phase 3 Study of Combination Antineoplaston Therapy [Antineoplastons A10 (Atengenal) and AS2-1 (Astugenal)] Plus Radiation Therapy vs. Radiation Therapy Only in Subjects With Newly Diagnosed Diffuse, Intrinsic, Brainstem Glioma
Brief Title: Study of Antineoplaston Therapy + Radiation vs. Radiation Only in Diffuse, Intrinsic, Brainstem Glioma
Acronym: DIPG
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRI-BT-52
Record Dates: First submitted 2016-08-09; First posted 2016-09-01 (Estimated); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Brain Stem Glioma
Keywords: Diffuse, intrinsic brain stem glioma; Antineoplaston therapy; Radiation
MeSH Terms: interventions — Radiation; antineoplaston A10

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Radiation (Experimental): Study subjects receive a single daily radiation fraction of 180cGy, 5 days a week for 6 weeks overall, to a total radiation dose of 5400cGy.
  Interventions: Radiation: Radiation
- Antineoplaston therapy + Radiation (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for 104 weeks. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached. Study subjects also receive a single daily radiation fraction of 180cGy, 5 days a week for 6 weeks overall, to a total radiation dose of 5400cGy.
  Interventions: Radiation: Radiation; Drug: Atengenal; Drug: Astugenal

INTERVENTIONS:
Radiation: Radiation — Subjects ≥ 3 years of age with a diffuse, intrinsic brain stem glioma will receive radiation.
Drug: Atengenal — Subjects ≥ 3 years of age with a diffuse, intrinsic brain stem glioma will receive Atengenal in combination with Astugenal (Antineoplaston therapy) and radiation
  Other Names: A10
  Arms: Antineoplaston therapy + Radiation
Drug: Astugenal — Subjects ≥ 3 years of age with a diffuse, intrinsic brain stem glioma will receive Astugenal in combination with Atengenal (Antineoplaston therapy) and radiation
  Other Names: AS2-1
  Arms: Antineoplaston therapy + Radiation

SUMMARY:
Patients ≥ 3 years of age with newly-diagnosed, diffuse, intrinsic pontine glioma will be enrolled in this study. However, the primary objectives of this study are to 1) compare overall survival, the time from randomization to death from any cause, for study subjects 3-21 years of age with newly-diagnosed, diffuse, intrinsic pontine glioma who receive Antineoplaston therapy (Atengenal + Astugenal) + radiation therapy vs. radiation therapy alone and 2) describe the toxicity profile (all subjects) for Antineoplaston therapy + radiation therapy vs. radiation therapy alone.

A secondary objective is to compare progression-free survival for study subjects 3-21 years of age with newly-diagnosed, diffuse, intrinsic pontine glioma treated with Antineoplaston therapy + radiation therapy vs. radiation therapy alone.

DETAILED DESCRIPTION:
This is a randomized Phase 3 protocol study of Antineoplaston therapy + radiation therapy vs. radiation therapy alone in subjects ≥ 3 years of age with newly-diagnosed, diffuse, intrinsic pontine glioma. In those subjects randomized to Antineoplaston therapy + radiation therapy, Antineoplaston therapy is administered for 104 weeks while radiation therapy commences on day one of Antineoplaston therapy and continues for 6 weeks. Subjects continue on Antineoplaston therapy if an objective response or stable disease is achieved during therapy and are maintained on Antineoplaston therapy to the end of the protocol study unless they develop progressive disease. Subjects randomized to radiation therapy alone receive 6 weeks of radiation therapy.

Exploratory objectives are to compare the following in the two treatment arms: 1) overall survival for study subjects ≥ 21 years of age; 2) progression-free survival for subjects ≥ 21 years of age; 3) objective response, complete response, partial response, and progressive disease rates, based on the enhancing portion of the tumor, for all subjects, using bidimentional measurement of tumor; 4) objective response, complete response, partial response, and progressive disease rates, for all subjects with non-enhancing tumors, using unidimentional measurement of tumor; and 5) objective response, complete response, partial response, and progressive disease rates, based on the enhancing + non-enhancing portions of the tumor, for all subjects, using unidimentional measurement of tumor.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Diffuse, Intrinsic Pontine Glioma as defined by the following criteria are eligible:

  * A characteristic MRI appearance, including variable contrast enhancement after gadolinium administration, diffuse T2/FLAIR signal, and involvement of more than 50% of the pons.
  * Confirmation of anaplastic glioma (i.e., oligodendroglioma, astrocytoma, oligoastrocytoma) or GBM histology if there is less than 50% involvement of the pons.
* Screening evaluation requires a MRI performed within 14 days prior to the start of ANP therapy. Study subjects must be on a fixed dose of steroids for at least five days prior to the screening MRI. If the steroid dose is changed between the date of imaging and the start of treatment, a new baseline MRI is required. All MRIs must be performed at an accredited radiology center. All MRIs should include at a minimum: T1-weighted images pre/post gadolinium administration, fluid attenuated inversion recovery (FLAIR), and T-2 weighted images.
* Subjects 3-21 years of age must have a clinical history of disease of less than 6 months and at least two of the following clinical findings: cranial nerve deficit, long tract signs (i.e. hemiparesis) and ataxia are eligible. Subjects > 21 years of age do not need to meet these criteria.
* Subjects must be ≥ 3 years of age. RT is not recommended for subjects less than 3 years of age.
* Subjects ≤ 16 years of age with a Lansky performance status of > 40 are eligible. Subjects > 16 years of age with a Karnofsky performance status of > 40 are eligible.
* Subjects with organ and marrow function (as defined below) are eligible.

  * Hemoglobin ≥ 9 g/dL
  * Leukocytes > 2000/mm3
  * Absolute neutrophil count >1,000/ mm3
  * Serum Na+ ≤ 150 mmol/L
  * Serum K+ ≤ 5.5 mmol/L
  * Serum creatinine ≤ 1.5 times institutional upper limit
  * Platelets >50,000/ mm3
  * Total bilirubin < 2.5 mg/dL
  * AST (SGOT) / ALT (SGPT) <5 times institutional upper limit
* At the recommended therapeutic dose, the effects of ANP therapy on the developing human fetus are unknown. For this reason, women of child-bearing potential who agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to protocol study entry and for the duration of the protocol study are eligible. Should a woman become pregnant or suspect she is pregnant while participating in this protocol study, she will inform her treating physician immediately.
* Subjects, parents, and/or guardians who are able to understand a written informed consent document, and are willing to sign it, are eligible.

Exclusion Criteria:

* No type of prior therapy, including other investigational agents, is allowable. A prior diagnostic biopsy or surgical shunt for hydrocephalus is permitted.
* Subjects with disseminated disease, multicentric tumors, leptomeningeal disease, or the history of retrotumoral bleeding are not eligible. The screening / baseline MRI includes the spinal cord to rule out leptomeningeal disease.
* Subjects with a known history of ganglioglioma are not eligible.
* Subjects with a current diagnosis or family history of neurofibromatosis I or II are not eligible. - Subjects with a current diagnosis or family history of neurofibromatosis are not eligible.
* Subjects with an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled hypertension despite maximal medical management (three supine blood pressure measurements ≥ 150/99 taken at least one hour apart) or psychiatric illness/social situations that would limit compliance with protocol study requirements are not eligible.
* Subjects with a history of New York Heart Association Class II congestive heart failure are not eligible.
* Pregnant women are not eligible because the teratogenic and abortifacient effects of ANP therapy in humans are unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to the mother receiving ANP therapy, breastfeeding is discontinued if the mother receives ANP therapy.

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Percentage of Participants Who Survived (Overall Survival) | 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
  The Kaplan-Meier nonparametric method is used to evaluate overall survival in the two therapy groups. Survival difference is evaluated using a log-rank test, which compares the two therapy groups. A Cox proportional hazards model is used as a supportive analysis to assess the magnitude of difference between the two therapy groups. The median survival rate in the two therapy groups (and 95% confidence intervals) is evaluated. Hazard ratio and its 95% confidence interval are estimated.

SECONDARY OUTCOMES:
Change in Percentage of Participants Who Survived (Progression-free Survival) | 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
  The Kaplan-Meier nonparametric method is used to evaluate progression-free survival in the two therapy groups. Progression-free survival difference is evaluated using a log-rank test, which compares the two therapy groups. A Cox proportional hazards model is used as a supportive analysis to assess the magnitude of difference between the two therapy groups. The median progression-free survival rate in the two therapy groups (and 95% confidence intervals) is evaluated. Hazard ratio and its 95% confidence interval are estimated.analysis is provided.

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Study Chair — Burzynski Research Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burzynski SR, Janicki J, Burzynski G, Marszalek A. A Phase II Study of Antineoplastons A10 and AS2-1 in Patients with Brainstem Gliomas. The Report on Non-Diffuse Intrinsic Pontine Glioma (Protocol BT-11). Journal of Cancer Therapy 6:334-344,2015. doi: 10.4236/jct.2015.64036
- [Background] Burzynski SR, Janicki TJ, Burzynski GS, Marszalek A. The response and survival of children with recurrent diffuse intrinsic pontine glioma based on phase II study of antineoplastons A10 and AS2-1 in patients with brainstem glioma. Childs Nerv Syst. 2014 Dec;30(12):2051-61. doi: 10.1007/s00381-014-2401-z. Epub 2014 Apr 10. PMID 24718705
- [Background] Burzynski SR. Recent clinical trials in diffuse intrinsic brainstem glioma. Cancer Therapy 5:379-390, 2007. Epub 2007 Nov
- [Background] Burzynski SR, Janicki TJ, Weaver RA, Burzynski B. Targeted therapy with antineoplastons A10 and AS2-1 of high-grade, recurrent, and progressive brainstem glioma. Integr Cancer Ther. 2006 Mar;5(1):40-7. doi: 10.1177/1534735405285380. PMID 16484713
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com